CLINICAL TRIAL: NCT03987009
Title: Do the Head-elevated Position and the Use of a Videolaryngoscope Facilitate Orotracheal Intubation in a Patient Population Without Predictable Difficulty of Intubation
Acronym: HELP-VDL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Discontinuation of DM production by the manufacturer leading to recruitment difficulties in the centers.
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017011F
Record Dates: First submitted 2019-06-07; First posted 2019-06-14 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Without RAMP and without video (Experimental): Sniffing position and a standard Macintosh laryngoscope
  Interventions: Device: Without RAMP and without video
- With RAMP and with video (Experimental): Ramped position and a McGrath Mac videolaryngoscope
  Interventions: Device: With RAMP and with video
- Without RAMP and with video (Experimental): Sniffing position and a McGrath Mac videolaryngoscope
  Interventions: Device: Without RAMP and with video
- With RAMP and without video (Experimental): Ramped position and a standard Macintosh laryngoscope
  Interventions: Device: With RAMP and without video

INTERVENTIONS:
Device: Without RAMP and without video — Intubation with video-laryngoscope McGrath without use of the video feature and patient positioning without RAMP device
  Arms: Without RAMP and without video
Device: With RAMP and with video — Intubation with video-laryngoscope McGrath with use of the video feature and patient positioning with RAMP device
  Arms: With RAMP and with video
Device: Without RAMP and with video — Intubation with video-laryngoscope McGrath with use of the video feature and patient positioning without RAMP device
  Arms: Without RAMP and with video
Device: With RAMP and without video — Intubation with video-laryngoscope McGrath without use of the video feature and patient positioning with RAMP device
  Arms: With RAMP and without video

SUMMARY:
The main hypothesis of this study is that there is a synergy between the use of the HELP position and the use of a McGrath® Mac videolaryngoscope to facilitate tracheal intubation during anesthesia.

The HELP position is the patient positioning on the AirPal RAMP, the two cushions inflated, bringing the external auditory canal to the same level as the sus-sternal notch.

DETAILED DESCRIPTION:
Airway management remains an important determinant of morbidity and mortality in anesthesia, despite progress in recognizing factors of difficult mask ventilation and intubation. Many recommendations have been published regarding the practice of intubation in anesthesia. Our study focuses on two topics which remain under discussion: the position of the patient's head and the use of a videolaryngoscope.

As to patient's head position, most anesthesiologists place the patient in the sniffing position (supine torso with neck flexed forward, and head extended), a position denominated "sniffing"by analogy to that adopted to smell a perfume. However, Adnet et al. questioned this position based on magnetic resonance imaging of eight healthy young volunteers positioned either with their heads in a neutral position or in extension, or with their heads and necks on a pillow. They showed that the sniffing position does not allow the alignment of the three important axes (mouth, pharynx and larynx) in awake patients with normal airway anatomy [1]. The "Head Elevated Laryngoscopic position" (HELP), with a raise of the head and neck so that "An imaginary horizontal line should connect the patient's sternal notch with the external auditory meatus" [2] facilitates the alignment of the pharyngeal, laryngeal, and oral axes of the airway during difficult laryngoscopy [3].

As to videolaryngoscopy, there is no doubt that it is a major advance in airway management. A recent Cochrane Systematic Review concluded that videolaryngoscopy increased easy laryngeal views and reduced difficult views and intubation difficulty [4]. However, its place is still debated: first line or rescue in case of suspected difficult airway. Its systematic use means discarding the standard Macintosh laryngoscope [5] which is not supported by clinical studies, in particular those of Wallace et al. [6] and of Thion et al. [7].

In the present randomized study we will study a combination of two factors in tracheal intubation on patients without suspected airways abnormalities: position (sniffing or HELP) and a McGrath laryngoscope (with or without video). This leads to four groups, A: sniffing position plus McGrath Mac videolaryngoscope with its screen deactivated so as to mimic a plain laryngoscope (R-V-), B: HELP plus McGrath Mac videolaryngoscope with a deactivated video screen (R+V-), C: sniffing position plus a McGrath Mac videolaryngoscope with an activated video screen (R-V+), D: HELP plus a McGrath Mac videolaryngoscope with it video screen activated (R+V+). This protocol allows using the same type of laryngoscope in all cases.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 89 years old
* Scheduled for elective surgical procedures
* Requiring oro-tracheal intubation for general anesthesia
* Having a telephone and agreeing to communicate their phone number in case of ambulatory surgery
* Having signed an informed consent form
* Benefiting from a social insurance

Exclusion Criteria:

* Pregnant or breast-feeding women
* Patients with an anticipated difficult mask ventilation or an anticipated difficult intubation (Arné's score ≥ 11)
* Patients scheduled for a surgical procedure involving the mouth or the upper airway
* Patients requiring a rapid induction sequence, the use of a double-lumen tube
* Patients having a contra-indication to one of the drug administered by the protocol

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
Proportion of oro-tracheal intubations for which it is necessary to use the assistance of a third party required by the operator | 30 minutes
  Intubation is video and audio recorded. The number of people nedeed is determined from the audio/video recording a posteriori by two independent evaluators

SECONDARY OUTCOMES:
Time to perform the intubation | 30 minutes
  Based on the video recording: from the passage the incisors to the third capnogram
First intubation succes rate | 30 minutes
  Defined by repositioning of the videolaryngoscope blade in the patient's mouth
Assessment of the Quality of visualization of the glottis | 30 minutes
  It is appreciated in real time by score of Cormak and Lehane modified by Yentis : from Grade 1 (glottis seen in totality) to Grade 4 (glottis hidden by epiglottis and tongue)
Assessment of the Percentage of the opening of the glottic orifice | 30 minutes
  It is appreciated in real time POGO (Percentage of Opening of the Glottic orifice) score : from 0% (opening not visible) to 100% (all of the opening is visible)
Assessment of quality of intubation with use of alternative techniques | 30 minutes
  Determined a posteriori from the video recording analysis
Occurrence of esophageal intubation | 30 minutes
  Reported in real time by the operator during the video / audio recording
Number of tracheal intubation failure | 30 minutes
  Number of tracheal intubation failure reported by the operator during the video / audio recording. Can be determined a posteriori from the video / audio recording.
Incidence of arterial oxygen desaturation (SpO2 < 92%) | 30 minutes
  Valued in real time and reported by the operator during the video / audio recording.
Perception of difficulty in intubation | 30 minutes
  Evaluation in real time based on a scale betwwen zero ( no difficulty) to ten (extremely difficult)
Cooperation of the various members of the anesthesia team | 30 minutes
  Determined from the video / audio recording using Kraus Scale to evaluate cooperation and non-cooperation behaviors within the team. Positive rating: scale from 0 (never reported by the obsever) to 4 (obvious to the obsever). Negative rating: scale from 0 (nerver reported by the observer) to 4 (obvious most of the time for the observer)
Evolution of Blood pressure | 30 minutes
  Blood pressure is monitored before the induction, before and after intubation.
Evolution of Heart beat | 30 minutes
  Heart beat is monitored before the induction, before and after intubation.
Evaluation of frequency of intubation complications | 24 hours
  Number of events of Sore throat and voice change evaluated during postoperative visit on day 1 of the surgery
Evaluation of severity of intubation complications | 24 hours
  Severity is evaluated during postoperative visit on day 1 of the surgery with 2 questions to the patient about his/her sore throat and voice change

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Le Guen, MD, Principal Investigator — Hôpital Foch
Locations (5):
- France (5):
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Hôpital Saint-Joseph, Paris
  - Institut Mutualiste Montsouris, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: Yes
Data will be available in the Dryad repository.
Supporting Information: Analytic Code
Time Frame: After publication in a peer-review journal. No limit in time
Access Criteria: No criteria
URL: https://datadryad.org/stash

REFERENCES:
- [Derived] Le Guen M, Coppere Z, Dufour G, Ouattara J, Trichereau J, Fischler M. HELP-VDL: study protocol for a multicentre, open, randomised, controlled clinical trial comparing the use of the head-elevated laryngoscopy position and the use of a videolaryngoscope to facilitate orotracheal intubation in a patient population without predictable difficulty of intubation. BMJ Open. 2020 Jul 8;10(7):e036570. doi: 10.1136/bmjopen-2019-036570. PMID 32641332